CLINICAL TRIAL: NCT02998099
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, PARALLEL-GROUP SINGLE-DOSE STUDY TO ESTIMATE THE EFFECT OF AGE ON THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF INTRAVENOUS RIVIPANSEL (PF-06460031)
Brief Title: A Study to Evaluate the Effect of Age on the Pharmacokinetics, Safety and Tolerability of IV Rivipansel.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B5201004
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Rivipansel
MeSH Terms: interventions — rivipansel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aged 18-45 years (Experimental): A single dose of IV rivipansel over 20 minutes.
  Interventions: Drug: Rivipansel
- Aged 65 and older (Experimental): A single dose of IV rivipansel over 20 minutes.
  Interventions: Drug: Rivipansel

INTERVENTIONS:
Drug: Rivipansel — A single dose of IV rivipansel over 20 minutes.
  Other Names: GMI-1070

SUMMARY:
The purpose of this study is to evaluate the effect of age on PK, safety and tolerability of IV rivipansel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential or healthy male subjects who are between the ages of 18-45 years or 65 years of age or older.
* Body mass index (BMI) of 17.5 to 40 kg/m2

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Pregnant females; breastfeeding female subjects; male subjects with partners currently pregnant
* Treatment with another investigational drug within 30 days or 5 half-lives preceding the dose of study medication
* Blood donation within 60 days prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time 0 extrapolated to infinite time or area under the plasma concentration-time from time 0 to time of the last quantifiable concentration as data permit. | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48 and 72 hours following single dose administration of IV rivipansel
Clearance (CL) | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48 and 72 hours following single dose administration of rivipansel.

SECONDARY OUTCOMES:
Area under the plasma concentration-time profile from time 0 to time of last quantifiable concentration | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48 and 72 hours following single dose administration of rivipansel.
Maximum plasma concentration | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48 and 72 hours following single dose administration of rivipansel.
Mean elimination half-life | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48 and 72 hours following single dose administration of rivipansel.
Volume of distribution at steady state | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48 and 72 hours following single dose administration of rivipansel.
Physical examination | Baseline up to 72 hours
Assessment of adverse events | Baseline up to 28 days
Assessment of 12-lead electrocardiogram | Baseline up to 72 hours
Assessment of vital signs | Baseline up to 72 hours
Assessment of laboratory tests | Baseline up to 72 hours

OTHER OUTCOMES:
Banked Biospecimen | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No